CLINICAL TRIAL: NCT00672074
Title: A Phase II, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety and Efficacy of Ipamorelin Compared to Placebo for the Management of Post-Operative Ileus in Patients
Brief Title: Safety and Efficacy of Ipamorelin for Management of Post-Operative Ileus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-IPAM-201
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Ileus
Keywords: Postoperative Ileus
MeSH Terms: conditions — Ileus | interventions — ipamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Ipamorelin (Active Comparator)
  Interventions: Drug: Ipamorelin
- 2 Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ipamorelin — IV
  Other Names: ST
  Arms: 1 Ipamorelin
Drug: placebo — IV
  Other Names: ST
  Arms: 2 Placebo

SUMMARY:
The purpose of this study is to determine if ipamorelin is safe and effective in the management of post-operative ileus.

DETAILED DESCRIPTION:
The safety and efficacy of ipamorelin in the management of post-operative ileus

ELIGIBILITY:
Inclusion Criteria:

* willing to comply with protocol
* undergoing bowel resection surgery
* ASA Class I-III
* Females must not be pregnant
* Body weight 40-150 kg

Exclusion Criteria:

* mentally incompetent or unable to provide informed consent
* clinically unstable
* significant liver disease
* clinically significant lab or EKG abnormalities
* alcohol or illicit drug abuse
* history of or current surgery that would prevent proper evaluation of safety or efficacy of drug

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Recovery of GI function | Until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Allen, Study Director — Helsinn Therapeutics (U.S.), Inc
Locations (19):
- United States (19):
  - USC/Norris Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Palo Alto Veterans Hospital, Palo Alto, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver VA Hospital, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Cleveland Clinic of Weston, Weston, Florida
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - UMass Memorial Healthcare, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Barnes Jewish Hospital, St Louis, Missouri
  - Stony Brook University Medical Center, Stony Brook, New York
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Pennsylvania State University, Hershey, Pennsylvania
  - St. Joseph Hospital, Tacoma, Washington

REFERENCES:
- [Derived] Beck DE, Sweeney WB, McCarter MD; Ipamorelin 201 Study Group. Prospective, randomized, controlled, proof-of-concept study of the Ghrelin mimetic ipamorelin for the management of postoperative ileus in bowel resection patients. Int J Colorectal Dis. 2014 Dec;29(12):1527-34. doi: 10.1007/s00384-014-2030-8. Epub 2014 Oct 21. PMID 25331030